CLINICAL TRIAL: NCT02405377
Title: Chinese People's Liberation Army General Hospital
Brief Title: Central Venous Pressure Guided Hydration Prevention for Contrast-Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, Attending doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14KMM02
Record Dates: First submitted 2015-03-23; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Cardio-Renal Syndrome
Keywords: contrast-induced nephropathy; hydration; Percutaneous coronary intervention
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — iodixanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVP guided hydration (Experimental): The fluid rate was adjusted according to the CVP dynamically
  Interventions: Procedure: hydration; Drug: Visipaque; Drug: 0.9% sodium chloride ﬂuid administration; Device: 5-French catheter
- Control (Active Comparator): The control group was hydrated at 1 mL/kg per h.
  Interventions: Procedure: hydration; Drug: Visipaque; Drug: 0.9% sodium chloride ﬂuid administration

INTERVENTIONS:
Procedure: hydration — Before the coronary procedures, investigators used the same 0.9% sodium chloride for hydration in all patients. Investigator monitored the central venous pressure (CVP) by placing an 5-French catheter in the jugular vein in the intervention group, and administration fluid rate was adjusted according to the CVP as follows: 3 ml/kg/h for CVP lower than 6 mmHg, 1.5 ml/kg/h for pressure of 6-12 mmHg, and 1ml/kg/h for pressure higher than 12 mmHg. The control group was hydrated with 0.9% sodium chloride at 1 ml/kg/h, continued for the duration of 12 h post-procedure in both groups. Thus, both study groups received intravenous fluids for the same duration but at different rates. All study participants received intra-arterial Visipaque(320 mg I/ml; GE Healthcare) iso-osmolar contrast medium.
Drug: Visipaque — All study participants received intra-arterial (320 mg I/ml; GE Healthcare)
Drug: 0.9% sodium chloride ﬂuid administration
Device: 5-French catheter
  Arms: CVP guided hydration

SUMMARY:
Patients at moderate and high risk for contrast induced nephropathy (CIN) should receive sufficient hydration before application of contrast to prevent CIN, but hydration could obviously increase the preload for congestive heart failure (CHF) patients. It is important to make an individual hydration protocol for patients with dysfunction of heart and renal to reduce the incidence rate of CIN. This prospective, randomized, double-blind, comparative clinical trial randomly selected 264 patients with estimated glomerular filtration rate, (eGFR) <60 ml/min per 1.73 m2 and CHF undergoing coronary angiography to receive either the convention hydration (n=132) or the central venous pressure (CVP) guided hydration (n=132).

DETAILED DESCRIPTION:
Investigators enrolled 264 patients from February 2014 to February 2015, the principal inclusion criterion included CHF: left ventricular eject fraction (LVEF) <= 50%; moderate to severe CKD was diagnosed as an eGFR 15 to 59 mL/min per 1.73 m2, calculated via the abbreviated Modification of Diet in Renal Disease (MDRD) study equation from SCr obtained within 72 hours of enrollment, patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions. We randomly assigned eligible patients in a 1:1 ratio to either CVP guided therapy or a standard hydration administration protocol. Investigators used the same fluid type commercially available 0.9% sodium chloride in all patients. Investigators monitored the CVP by placing an 5-French catheter in the jugular vein. Investigators recorded the CVP with commercially available haemodynamic monitoring software. In the CVP guided group the fluid rate was adjusted according to the CVP as follows: 3 mL/kg/h for CVP lower than 6 mmHg, 1.5 mL/kg/h for pressure of 6-12 mmHg, and 1mL/kg/h for pressure higher than 12 mmHg. The control group was hydrated at 1 mL/kg per h. The fluid rate was set at the start of the procedure (before contrast exposure). Thus, both study groups received intravenous fluids for the same duration but at different rates. All study participants received intra-arterial Visipaque(320 mg I/ml; GE Healthcare) iso-osmolar contrast medium.

Primary end point of the study was the incidence of CIN: The median peak increase in serum creatinine concentration between day 0 (when contrast was administered) and day 7. Definition of CIN was an absolute increase in serum creatinine (SCr) >0.5 mg/dl or a relative increase >25% compared to baseline SCr. Definition of non-Q-wave myocardial infarction was a creatine kinase-myocardial band enzyme elevation 3 times the upper normal value without new Q waves on the electrocardiogram. Definition of Q-wave myocardial infarction was presence of new pathologic Q waves on an electrocardiogram in conjunction with an elevation in creatine kinase greater than 3 times the normal value. All adverse clinical events as well as study end points were monitored and adjudicated by the independent event committee. Each patient was contacted in every week after administration of the contrast, investigated if dialysis or main cardiovascular events (myocardial infarction,acute heart failure and death), and record any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. congestive heart failure: objective evidences for decreased left ventricular eject fraction (LVEF) <= 50%;
2. moderate to severe chronic kidney disease was defined as an eGFR 15 to 59 mL/min per 1.73 m2, calculated via the abbreviated Modification of Diet in Renal Disease (MDRD) study equation from SCr obtained within 72 hours of enrollment;
3. patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions.

Exclusion Criteria:

1. hemodialysis-dependent patients;
2. complicated with severe short-term progressive disease;
3. Patients < 18 years;
4. pregnancy;
5. emergency cardiac catheterisation (eg, primary percutaneous coronary intervention for ST-segment elevation myocardial infarction);
6. exposure to radiographic contrast media within the previous 7 days;
7. acute decompensated heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy postoperation | 7 days
  a peak serum creatinine increase of either 0.5 mg/dl or 25% from day 0 through day 7

SECONDARY OUTCOMES:
Composite measure of dialysis or main cardiovascular events | 90 days
  dialysis, myocardial infarction, heart failure and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Dai Yun Chen, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Schilp J, de Blok C, Langelaan M, Spreeuwenberg P, Wagner C. Guideline adherence for identification and hydration of high-risk hospital patients for contrast-induced nephropathy. BMC Nephrol. 2014 Jan 6;15:2. doi: 10.1186/1471-2369-15-2. PMID 24393347
- [Background] Balemans CE, Reichert LJ, van Schelven BI, van den Brand JA, Wetzels JF. Epidemiology of contrast material-induced nephropathy in the era of hydration. Radiology. 2012 Jun;263(3):706-13. doi: 10.1148/radiol.12111667. Epub 2012 Apr 24. PMID 22535561
- [Background] Marenzi G, Ferrari C, Marana I, Assanelli E, De Metrio M, Teruzzi G, Veglia F, Fabbiocchi F, Montorsi P, Bartorelli AL. Prevention of contrast nephropathy by furosemide with matched hydration: the MYTHOS (Induced Diuresis With Matched Hydration Compared to Standard Hydration for Contrast Induced Nephropathy Prevention) trial. JACC Cardiovasc Interv. 2012 Jan;5(1):90-7. doi: 10.1016/j.jcin.2011.08.017. PMID 22230154
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Torigoe K, Tamura A, Watanabe T, Kadota J. 20-Hour preprocedural hydration is not superior to 5-hour preprocedural hydration in the prevention of contrast-induced increases in serum creatinine and cystatin C. Int J Cardiol. 2013 Sep 1;167(5):2200-3. doi: 10.1016/j.ijcard.2012.05.122. Epub 2012 Jun 19. PMID 22717305
- [Background] Duan N, Zhao J, Li Z, Dong P, Wang S, Zhao Y, Wang L, Wang H. Furosemide with saline hydration for prevention of contrast-induced nephropathy in patients undergoing coronary angiography: a meta-analysis of randomized controlled trials. Med Sci Monit. 2015 Jan 23;21:292-7. doi: 10.12659/MSM.892446. PMID 25613017
- [Result] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Derived] Qian G, Fu Z, Guo J, Cao F, Chen Y. Prevention of Contrast-Induced Nephropathy by Central Venous Pressure-Guided Fluid Administration in Chronic Kidney Disease and Congestive Heart Failure Patients. JACC Cardiovasc Interv. 2016 Jan 11;9(1):89-96. doi: 10.1016/j.jcin.2015.09.026. Epub 2015 Dec 9. PMID 26685074